CLINICAL TRIAL: NCT06884085
Title: An Open-label, Randomized, Single-dose, 2-sequence, 2-period, Crossover Study to Evaluate the Safety and Pharmacokinetics of AD-227 Compared to Co-administration of AD-227A and AD-227B in Healthy Adult Volunteers Under Fasting Conditions
Brief Title: A Study to Compare to PK Characteristics and Safety Profiles Between AD-227 and Co-administration of AD-227A and AD-227B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AD-227BE-02
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Primary Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (RT) (Experimental): Period 1: Reference (Co-administration of AD-227A and AD-227B), Period 2: Test (AD-227)
  Interventions: Drug: Co-administration of AD-227A and AD-227B; Drug: Administration of AD-227
- Sequene B (TR) (Experimental): Period 1: Test (AD-227), Period 2: Reference (Co-administration of AD-227A and AD-227B)
  Interventions: Drug: Co-administration of AD-227A and AD-227B; Drug: Administration of AD-227

INTERVENTIONS:
Drug: Co-administration of AD-227A and AD-227B — Co-administration of AD-227A 1Tab. and AD-227B 1Tab., Per Oral
Drug: Administration of AD-227 — Administration of AD-227 1Tab., Per Oral

SUMMARY:
Primary endpoint of this study is to evaluate the pharmacokinetic characteristics of AD-227 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body weight equal to or greater than 50kg (Female 45kg) and Body mass index (BMI) between 18.0 kg/m2 and 30.0 kg/m2 at the time of screening visit
* The Age equal to or greater than 19 in healthy volunteers at the time of screening visit

Exclusion Criteria:

* Participation in another clinical study with an investigational drug within the 6 months from scheduled first administration
* Other exclusions applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-07-12 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Maximum concentration of drug in plasma (Cmax) | pre-dose (0hour) to 72hours
  Cmax of AD-227
Area under the plasma concentration-time curve during dosing interval (AUCt) | pre-dose (0hour) to 72hours
  AUCt of AD-227

CONTACTS AND LOCATIONS:
Locations (1):
- Central Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No